CLINICAL TRIAL: NCT04693832
Title: Trakya University, Scientific Research Projects Unit
Brief Title: The Effect of Using Interactive Mobile Application for the Management of Chemotherapy- Induced Nausea and Vomiting in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Remziye Semerci, Research Assistant, Trakya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Remziye Semerci
Record Dates: First submitted 2020-12-23; First posted 2021-01-05 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Oncology; Nausea and Vomiting Chemotherapy-Induced; Pediatric Cancer; Mobile Application
MeSH Terms: conditions — Neoplasms; Nausea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5inD (Experimental): All children receive routine antiemetic therapy before chemotherapy. Children in the experimental group will use the interactive mobile application (5inD) for seven days from the first day of chemotherapy. The games in this application will help distract their attention and manage their nausea and vomiting.
  Interventions: Device: 5inD
- Control group (No Intervention): All children receive routine antiemetic therapy before chemotherapy.

INTERVENTIONS:
Device: 5inD — Interactive Mobile Application which is includes five different game (mandala, puzzle, tetris, music, breath exercise)
  Arms: 5inD

SUMMARY:
The aim of this study was to develop an interactive mobile application and to investigate the effect of this application on the management of nausea and vomiting symptoms by using it during chemotherapy treatment.

DETAILED DESCRIPTION:
Intensive chemotherapy protocols are the most commonly used treatments in childhood cancers. While these protocols increase recovery rates, they may also cause some undesirable side effects. Nausea and vomiting are one of the most common toxic side effects associated with chemotherapy. The aim of this study was to develop an interactive mobile application and to investigate the effect of this application on the management of nausea and vomiting symptoms by using it during chemotherapy treatment.

The study will be conducted with 61 children between 8-18 years of age who received chemotherapy in the Pediatric Hematology-Oncology Clinic at Trakya University Health Research and Application Center. The study was planned as a randomized controlled study. Data will be collected with the "Information Form" and "Rhodes Adapted Rhodes Nausea and Vomiting Scale for Children". The interactive mobile application will be downloaded to the phones of the experimental group and this device will be used from the first chemotherapy day to the seventh day. While the experimental group evaluates their nausea and vomiting via mobile application twice a day, every 12 hours for one week, the control group will record their nausea and vomiting experiences in the "Nausea and Vomiting Diary". While the experimental group will be able to use the mobile application which consists of diverting attention, routine control will be applied to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Taking chemotherapy treatment,
* To be in the age range of 8-18,
* Volunteering to participate in research,
* Having the first course of chemotherapy,

Exclusion Criteria:

* Having a mental problem,
* Absence of vision, hearing and speech problems,
* Absence of problems with the gastrointestinal system,
* Being in the terminal period,
* Receiving sedation therapy,

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Adapted Rhodes Index of Nausea and Vomiting for Pediatrics | Both children and their mother's assess children's frequency of the nause and vomiting twice a day, every 12 hours during one week from the first chemotherap' day to the seventh day.
  The instrument consists of a series of 5 statements (rated 0-4) for each of the 6 items representing the child's perceptions of the frequency of, duration of, and distress from nausea, and the frequency of, amount of, and distress from vomiting within the past 12 hours.
  The ARINV includes 6 items. The first 3 items on the scale question the frequency of, amount of, and distress from vomiting during the last 12 hours and the remaining 3 items question the frequency of, duration of, and distress from nausea. The possible minimum and maximum scores to be obtained from the nausea or vomiting part of the ARINV vary between 0 and 24 per day. The possible minimum and maximum scores to be obtained from the whole ARINV vary between 0 and 48 per day.
Information Form | Children and parents complete this form before the study.
  The information form developed by the researchers includes the socio-demographic characteristics of parents and children; mother's age, father's age, parents 'education level, parents' employment status, number of children, child's age, gender, time of diagnosis of the child, disease stage of the child, types of treatment received, the number of cycles. It consists of 20 questions.

CONTACTS AND LOCATIONS:
Locations (1):
- Trakya University, Edirne, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided